CLINICAL TRIAL: NCT02681250
Title: A Randomized Controlled Clinical Trial of Dental Implants in Titanium-zirconium Alloy
Brief Title: A Clinical Trial of Dental Implants in Titanium-zirconium Alloy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TiZir
Record Dates: First submitted 2016-02-01; First posted 2016-02-12 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Endosseous Dental Implant Failure
Keywords: Zirconium; Randomized Controlled Trial; Dental Implants; Dental Material; Titanium
MeSH Terms: interventions — titanium alloy (TiNb13Zr13); Titanium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium-zirconium (Experimental): Patients receiving titanium-zirconium implants
  Interventions: Procedure: Titanium-zirconium
- Titanium (Active Comparator): Patients receiving titanium implants
  Interventions: Procedure: Titanium

INTERVENTIONS:
Procedure: Titanium-zirconium — Titanium-zirconium implants will be installed according to the protocol earlier described in the detailed description.
  Other Names: Straumann Roxolid SLA
  Arms: Titanium-zirconium
Procedure: Titanium — Titanium implants will be installed according to the protocol earlier described in the detailed description.
  Other Names: Straumann SLA (Sand blasted, Large grit, Acid Etched)
  Arms: Titanium

SUMMARY:
A Randomized controlled Clinical trial which aim is to investigate the clinical outcome of dental implants in titanium-zirconium alloy compared to traditional titan-4 implants. The hypothesis is set to no difference in the clinical outcome for the two types of implants. Preliminary estimation of 96 patients needed. A pilot study will provide us with further data in order to more accurately specify the sample number."

DETAILED DESCRIPTION:
Background

Implants have been used for the purpose of replacing lost teeth since the 1960s. Since then, the treatment of edentulism with dental implants has been implemented in a large scale. The main reason for this is that research has shown that treatment with implants are very predictable in terms of implant survival. The accumulated knowledge, as seen from 15 and 20 year follow-ups, has been based on prerequisites that are not always followed today. One of them is that the implants used in the aforementioned studies are manufactured in titanium that has good rigidity and is used as the main implant material today. In addition, the studies have examined implants with a turned surface. This standard revised in the mid 1990s when a series of studies showed increased and accelerated osseous ingrowth of implants with a moderate raw surface that had been achieved by blasting. The related biological events describing this process have been described in detail in the literature.

Today, other materials are being explored as an alternative to the well documented implant material titanium with a focus on finding a material with higher stiffness combined with equivalent biological characteristics. A stiffer material theoretically gives possibilities for implants installations without bone augmentation in cases with reduced bone volumes.

An alternative implant material which has reached the clinic is titanium-zirconium alloy. It has been shown to have an increased rigidity in comparison with titanium and comparable biological characteristics but the documentation consists mainly of animal studies and short term clinical follow-up in the form of case-series. Since it has been demonstrated that the choice of implant material may influence osseointegration, it is necessary to evaluate the implants made of titanium-zirconium in a clinical controlled study with long-term follow-up in which the emphasis is put on the clinical outcome.

Aims

The aim of the study is to compare the clinical outcome of implants made of titanium-zirconium with a proven implants made of titanium.

The scientific question in this project is if there are differences in the clinical outcomes of an implant made of titanium and a corresponding implants in titanium-zirconium alloy.

Materials and Methods

Patients referred for implant treatment at the Department of Prosthodontics, Specialisttandvården Borås will be asked to participate in the study and provide written consent after review of delivered information sheet. Implants will be installed by two well experienced surgeons at Oral Maxillofacial Surgery att Borås Regional Hospital according to the protocol used for dental implant surgery and recommended by the manufacturer.

Two groups, matched for age and gender, will be defined after block randomisation for smoking. The test group will receive titanium-zirconium implants and the control group titanium implants. For a power of 80% and for p < 0.05, (SD = 1.66 according to previous studies, estimates made from 1 mm difference in margin bone level between the groups), the size of the groups has been defined as 44 patients per group. The investigators anticipate a loss of approximately 10% and therefore, the investigators have increased each patient group to 48 individuals. The data collection is completed when the number of patients has been reached.

The evaluation will involve no additional clinical or radiological examinations as compared to the usual procedures. Normally, this means examination and therapy planning, surgical examination, implant installation, impression, placement of prosthetic restoration, baseline X-ray, control/follow-up tightening of prosthetic screw/hygiene monitoring. No additional time or costs arises in connection with participation in the study, the cost of both groups are equivalent.

National guidelines will be followed regarding possible need of antibiotic prophylaxis. Registration will be done with regard to history of periodontal disease, smoking, medication, and implant position in the jaw.

The data collection will take place at four different times: in connection with the placement of the prosthetic construction (baseline) and after 1.3 and 5 years. Standard x-ray examinations will be carried out to check the marginal bone level which will take place through individualized x-ray holders that will be produced by impression material (Putty). Registration of pocket depth, bleeding on probing, amount of keratinized mucosa and measurements on x-ray will be done by the same person. Prosthetic complications and possible total implant loss will be registered.

The marginal bone level for each implant will be presented as the average of the mesial and distal bone level (primary outcome). The mean value of pocket depth will be recorded for each implant at a 4-point measurement. The hypothesis is to be tested with the independent samples t-test.

The impact of restoration distance from the bone level, the effect of implant type, margin bone level, bleeding on probing and pocket depth will be controlled using regression analysis. SPSS is used for statistical analysis.

The hypothesis is that there are no differences in the clinical outcomes between the two types of implants.

Potential benefits of the Project

The investigators can conclude that the materials are equivalent if there is no difference between implant types available. Since, titanium-zirconium alloy has a higher stiffness than titan, the investigators will be able to provide patients with thinner implant and thus costly and painful treatments to optimize the width of the bone in the installation area should be avoided.

From a social perspective, if it turns out that titan-zirconium have equal or better clinical performance than titanium, can unnecessary healthcare costs for surgery for modulation of the surgical site in the form of augmentation or sinus elevation associated with implant treatment should be avoided. If optimizing surgery can be avoided, this means even shorter therapy times and increased availability by the released health time which can be used to more quickly treat other patients as possible had standing in line for their treatment. Limits can be found in the study's applicability in general dentistry because all operations are carried out at specialist clinic in which case the patient clientele and the processor's level of expertise is not fully comparable with the general dentist.

Research ethical considerations

Treatment with dental implants in titanium is a known treatment that has helped to restore good chewing function for many patients and years all over the world and can be thought of as a safe treatment with high success rates. The study protocol calls for no difference in the x-ray examination or the surgical protocol as compared to the procedures followed in regular treatment basis. In previous studies, there is no listing of suspected allergy to titanium-zirconium alloy.

Patient information and storage of personal data in accordance with the recommendations of the Board of ethical review.

ELIGIBILITY:
Inclusion Criteria:

* All patients in need for implant treatment

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-02-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in bone loss measured on X-ray (mm) | Baseline and 1 year

SECONDARY OUTCOMES:
Change in bleeding on probing (Yes/No) | Baseline and 1 year
Change in amount of Clinical Mucosa (mm) | Baseline and 1 year
Change in Pocket depth (mm) | Baseline and 1 year
Change in Prosthetic Complications (Yes/No) | Baseline and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Bougas, PhD, Principal Investigator — Borås Regional Hospital
Locations (1):
- Specialisttandvården Borås, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branemark PI, Adell R, Breine U, Hansson BO, Lindstrom J, Ohlsson A. Intra-osseous anchorage of dental prostheses. I. Experimental studies. Scand J Plast Reconstr Surg. 1969;3(2):81-100. doi: 10.3109/02844316909036699. No abstract available. PMID 4924041
- [Background] Ekelund JA, Lindquist LW, Carlsson GE, Jemt T. Implant treatment in the edentulous mandible: a prospective study on Branemark system implants over more than 20 years. Int J Prosthodont. 2003 Nov-Dec;16(6):602-8. PMID 14714838
- [Background] Jemt T. Single implants in the anterior maxilla after 15 years of follow-up: comparison with central implants in the edentulous maxilla. Int J Prosthodont. 2008 Sep-Oct;21(5):400-8. PMID 18950060
- [Background] Jemt T, Ahlberg G, Henriksson K, Bondevik O. Changes of anterior clinical crown height in patients provided with single-implant restorations after more than 15 years of follow-up. Int J Prosthodont. 2006 Sep-Oct;19(5):455-61. PMID 17323723
- [Background] Wennerberg A, Albrektsson T, Andersson B. Bone tissue response to commercially pure titanium implants blasted with fine and coarse particles of aluminum oxide. Int J Oral Maxillofac Implants. 1996 Jan-Feb;11(1):38-45. PMID 8820121
- [Background] Wennerberg A, Albrektsson T, Johansson C, Andersson B. Experimental study of turned and grit-blasted screw-shaped implants with special emphasis on effects of blasting material and surface topography. Biomaterials. 1996 Jan;17(1):15-22. doi: 10.1016/0142-9612(96)80750-2. PMID 8962942
- [Background] Wennerberg A, Albrektsson T, Lausmaa J. Torque and histomorphometric evaluation of c.p. titanium screws blasted with 25- and 75-microns-sized particles of Al2O3. J Biomed Mater Res. 1996 Feb;30(2):251-60. doi: 10.1002/(SICI)1097-4636(199602)30:23.0.CO;2-P. PMID 9019491
- [Background] Berglundh T, Abrahamsson I, Lang NP, Lindhe J. De novo alveolar bone formation adjacent to endosseous implants. Clin Oral Implants Res. 2003 Jun;14(3):251-62. doi: 10.1034/j.1600-0501.2003.00972.x. PMID 12755774
- [Background] Bougas K, Jimbo R, Vandeweghe S, Hayashi M, Bryington M, Kozai Y, Schwartz-Filho HO, Tovar N, Adolfsson E, Ono D, Coelho PG, Wennerberg A. Bone apposition to laminin-1 coated implants: histologic and 3D evaluation. Int J Oral Maxillofac Surg. 2013 May;42(5):677-82. doi: 10.1016/j.ijom.2012.11.008. Epub 2012 Dec 8. PMID 23228694
- [Background] Kobayashi E, Matsumoto S, Doi H, Yoneyama T, Hamanaka H. Mechanical properties of the binary titanium-zirconium alloys and their potential for biomedical materials. J Biomed Mater Res. 1995 Aug;29(8):943-50. doi: 10.1002/jbm.820290805. PMID 7593037
- [Background] Gottlow J, Dard M, Kjellson F, Obrecht M, Sennerby L. Evaluation of a new titanium-zirconium dental implant: a biomechanical and histological comparative study in the mini pig. Clin Implant Dent Relat Res. 2012 Aug;14(4):538-45. doi: 10.1111/j.1708-8208.2010.00289.x. Epub 2010 Jun 25. PMID 20586785
- [Background] Wen B, Zhu F, Li Z, Zhang P, Lin X, Dard M. The osseointegration behavior of titanium-zirconium implants in ovariectomized rabbits. Clin Oral Implants Res. 2014 Jul;25(7):819-25. doi: 10.1111/clr.12141. Epub 2013 Feb 21. PMID 23432001
- [Background] Barter S, Stone P, Bragger U. A pilot study to evaluate the success and survival rate of titanium-zirconium implants in partially edentulous patients: results after 24 months of follow-up. Clin Oral Implants Res. 2012 Jul;23(7):873-81. doi: 10.1111/j.1600-0501.2011.02231.x. Epub 2011 Jun 24. PMID 21707752
- [Background] Benic GI, Gallucci GO, Mokti M, Hammerle CH, Weber HP, Jung RE. Titanium-zirconium narrow-diameter versus titanium regular-diameter implants for anterior and premolar single crowns: 1-year results of a randomized controlled clinical study. J Clin Periodontol. 2013 Nov;40(11):1052-61. doi: 10.1111/jcpe.12156. Epub 2013 Sep 8. PMID 24015975
- [Background] Nicolau P, Korostoff J, Ganeles J, Jackowski J, Krafft T, Neves M, Divi J, Rasse M, Guerra F, Fischer K. Immediate and early loading of chemically modified implants in posterior jaws: 3-year results from a prospective randomized multicenter study. Clin Implant Dent Relat Res. 2013 Aug;15(4):600-12. doi: 10.1111/j.1708-8208.2011.00418.x. Epub 2011 Dec 15. PMID 22171722
- [Background] Chrcanovic BR, Albrektsson T, Wennerberg A. Smoking and dental implants: A systematic review and meta-analysis. J Dent. 2015 May;43(5):487-98. doi: 10.1016/j.jdent.2015.03.003. Epub 2015 Mar 14. PMID 25778741
- [Background] Weber HP, Buser D, Fiorellini JP, Williams RC. Radiographic evaluation of crestal bone levels adjacent to nonsubmerged titanium implants. Clin Oral Implants Res. 1992 Dec;3(4):181-8. doi: 10.1034/j.1600-0501.1992.030405.x. PMID 1298433
- [Background] Hermann JS, Cochran DL, Nummikoski PV, Buser D. Crestal bone changes around titanium implants. A radiographic evaluation of unloaded nonsubmerged and submerged implants in the canine mandible. J Periodontol. 1997 Nov;68(11):1117-30. doi: 10.1902/jop.1997.68.11.1117. PMID 9407406